CLINICAL TRIAL: NCT04394169
Title: Early Care, Therapeutic Education, and Psychological Intervention for the Management of Post-intensive Care Syndrome and Chronic Pain After Coronavirus Disease 2019 Infection. Simple-blind, Controlled, Randomized Trial.
Brief Title: Early Care Program for the Management of Post-ICU Syndrome and Chronic Pain After COVID-19 Infection.
Acronym: PAIN-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, TOMAS MIGUEL CUÑAT LOPEZ, Collaborator Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HCB/2020/0549
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Post ICU Syndrome; Chronic Pain; Covid-19
Keywords: Covid-19; SARS-COV2; Critical Care; Post ICU Syndrome; Chronic Pain; Post-traumatic Stress Disorder; Quality of Life; Depressive Disorders; Anxiety disorders
MeSH Terms: conditions — Chronic Pain; COVID-19; Stress Disorders, Post-Traumatic; Depressive Disorder; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, single-blind, and single-center clinical trial that will include patients who have been admitted to intensive care of our hospital due to COVID-19 disease.
Who Masked: Investigator
Masking Description: Visits 1,2, and 3 will be carried out by an investigator with sufficient training in questionnaires. This investigator will not participate on the intervention or the evaluation of the results.
  The intervention will be performed by two researchers (Pain Physician and psychologist). This researcher will not participate in the questionnaire and basal data collection visits or results analysis.
  Researchers who analyze the results will not participate in the questionnaire and basal data collection or program intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The intervention is a program that includes early patient care, therapeutic education, and psychological intervention. It will be performed through three medical visits and a psychological intervention that requires seven face-to-face sessions.
  Interventions: Behavioral: Intervention program
- Standard care arm (No Intervention): Standard medical practice: patient follow-up is carried out by their referring physicians (primary care physicians or specialists) who are outside the study.

INTERVENTIONS:
Behavioral: Intervention program — Medical visits:
  There will be three medical visits stipulated as follows:
  * Visit 1 Intervention Group, four weeks after hospital discharge.
  * Visit 2 Intervention Group, eight weeks after hospital discharge.
  * Visit 3 Intervention Group, 18 weeks after hospital discharge.
  Components of visits:
  * Interview and physical examination.
  * Therapeutic education about the intensive care syndrome orally and with a specific document that will be delivered at the end of the visit.
  * Therapeutic education around pain. If the patient reports pain, a specific document will be prepared that will be delivered at the end of the visit.
  Psychological intervention:
  Inclusion criteria for psychological intervention: Patients with a score higher than 8 on the HAD (hospital anxiety and depression) test depression subscale.
  Description :
  The intervention protocol consists of 7 weekly sessions lasting one hour and a half. The intervention in depression is based on Rehm's model of self-control.
  Arms: Intervention arm

SUMMARY:
COVID-19 (coronavirus 2019) disease has led to a large number of hospital admissions, many of which require admission to intensive care (ICU).

Post-intensive care syndrome (PICS) is defined as deterioration or worsening of previous deterioration in the mental, physical or cognitive status that appears as a consequence of a critical illness and which persists after acute hospital care. Also, there is evidence that patients who survive a critical illness have a high prevalence of moderate to extreme chronic pain.

Patients with COVID-19 disease are an especially susceptible population to develop PICS due to acute respiratory distress syndrome (ARDS) survivors have significant long-term deterioration in mental, cognitive, and functional health.

This study hypothesis is that a specific care program based on early therapeutic education and psychological intervention improves the quality of life of patients at risk of developing PICS and chronic pain after COVID-19 disease.

DETAILED DESCRIPTION:
A randomized, controlled, and single-blind trial will be performed. Patients over 18 years who have been admitted to intensive care units with the diagnosis of COVID-19 disease at risk of presenting PICS will be recruited.

The study subjects will be divided into two arms, and the intervention program will be compared to the standard care clinical practice.

The program will consist of early care (first visit at one month of hospital discharge), therapeutic education on prevention and management of PICS and chronic pain during three medical visits in six months, and psychological treatment in patients at risk for emotional distress.

The main objective is to evaluate the impact of the program on health-related life quality at six months after hospital discharge.

The secondary objectives are:

1. To assess the health-related life quality at three months after hospital discharge.
2. To quantify the incidence of chronic pain, its characteristics, and the degree of functional limitation at three and six months after hospital discharge.
3. To quantify the incidence of anxiety and depression at three and six months after hospital discharge.
4. Quantify the incidence of post-traumatic stress syndrome at 3 and 6 months after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ICU due to COVID infection19.
* APACHE II score> 14 or ICU stay> 10 days or Duration of mechanical ventilation> 7 days or Acquired weakness in ICU or Delirium during ICU admission.
* Accept to participate in the study and sign informed consent.

Exclusion Criteria:

* Central Nervous System degenerative diseases. Examples: Alzheimer's disease, Amyotrophic lateral sclerosis, Lewy body dementia, Parkinson's disease, among others.
* Terminal illness: Definition according to the palliative care guide, Spanish Society for Palliative Care. "Advanced, progressive, and incurable disease with a lack of reasonable possibilities of specific treatment, with a life prognosis of less than 6 months.
* Insufficient understanding of the Spanish language.
* Patients in whom it would be difficult to complete follow-up.
* Not having informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Impact of intervention program on health-related quality of life (VAS) | Six months after discharge
  Health-related quality of life reported by the patient assessed through the visual analogue scale of the EQoL 5D/5L questionnaire at six months after discharge.
  [European quality of life 5 dimensions/5 levels ; from 0 (the worst imaginable health) to 100 (the best imaginable health) ]

SECONDARY OUTCOMES:
Impact of intervention program on health-related quality of life (VAS) | Three months after discharge.
  Health-related quality of life reported by the patient assessed through the visual analogue scale of the EQoL 5D / 5L questionnaire at three months after discharge.
  [European quality of life 5 dimensions/5 levels ; from 0 (the worst imaginable health) to 100 (the best imaginable health)]
Impact of intervention program on health-related quality of life (Index) | Three months after discharge
  Health-related quality of life reported by the patient assessed through health index of the EQoL 5D/5L questionnaire at three months after discharge.
  [European quality of life 5 dimensions/5 levels ; the questionnaire assesses quality of life in study participants according to 5 domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each scored according to a scale of 1 (no problems) to 5 (indicating extreme problems) and generating a 5-digit code corresponding to quality of life]
Impact of intervention program on health-related quality of life (Index) | Six months after discharge
  Health-related quality of life reported by the patient assessed through health index of the EQoL 5D/5L questionnaire at six months after discharge.
  [European quality of life 5 dimensions/5 levels ; the questionnaire assesses quality of life in study participants according to 5 domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each scored according to a scale of 1 (no problems) to 5 (indicating extreme problems) and generating a 5-digit code corresponding to quality of life]
Impact of intervention program on chronic pain (intensity) | Three and six months after discharge.
  Chronic pain intensity defined by BPI questionnaire (short version), at three and six months after discharge.
  [Brief pain inventory; A multidimensional questionnaire that evaluates pain intensity in the last 24 hours (worst, lowest, average) and current (right now). The questions are rated on a scale of 0 to 10, with 10 being the worst possible value. Subsequently, the average intensity score (BPI intensity score) is calculated.]
Impact of intervention program on chronic pain (limitation of daily activities) | Three and six months after discharge.
  Limitation of daily activities due to chronic pain, defined by BPI (short version), at three and six months after discharge.
  [Brief pain inventory; Multidimensional questionnaire that assesses the impact of pain on daily activities (general activity, encouragement, work, relationships with other people, sleep, enjoying life and the ability to walk). The questions are rated on a scale of 0 to 10, with 10 being the worst possible value. Subsequently, the mean score of the responses related to pain interference in activities (BPI interference score) is calculated.]
Impact of intervention program on chronic pain (Pain catastrophization) | Three and six months after discharge.
  Pain catastrophization assessed by Pain Catastrophizing Scale at three and six months after hospital discharge.
  [Pain Catastrophizing Scale; Consisting of 13 questions that explore the frequency of thoughts and feelings that the interviewees have in the presence of current or anticipated pain, which are grouped into three scoring subscales (magnification, rumination and defenselessness). Each question is rated on a 5-point scale (0: not at all; 4: all the time). Being the maximum total score of 52 points.]
Impact of intervention program on anxiety or depression incidence | Three and six months after discharge.
  Clinically significant anxiety or depression symptoms prevalence at three and six months, assessed by the HAD test.
  [hospital anxiety and depression test; 14 questions, with two subscales, one for anxiety and the other for depression, with seven items each, the maximum score is 21 for each subscale. The cut-off points from zero to seven imply the absence of clinically relevant anxiety and depression, from eight to ten symptoms that require consideration and from 11 to 21 reports the presence of relevant symptoms, with a very probable diagnosis of anxiety or depression.]
Impact of intervention on probable post-traumatic stress syndrome incidence | Three and six months after discharge.
  Probable post-traumatic stress syndrome prevalence at three and six months after discharge assessed by the DSM ( Diagnostic and Statistical Manual of Mental Disorders) V PTSD Checklist questionnaire (PCL-5)
  [PTSD Checklist questionnaire; It contains 20 questions that correspond to the DSM V PTSD (Post Traumatic Stress Disorder) criteria. Participants rated their symptoms on a scale of 0 (not at all), 1 (slightly), 2 (moderately), 3 (quite) to 4 (extremely), with a score ranging from 0 to 80. A total of the severity of the symptoms can be made, adding the score of each question (interval 0-80). The severity of each symptom can be evaluated, adding the score of the questions. The cut-off point to use for a provisional diagnosis of PTSD is 31 points.]

CONTACTS AND LOCATIONS:
Overall Officials: Antonio José Ojeda Niño, MD, Principal Investigator — Pain unit physician
Locations (1):
- Tomás Cuñat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Mao L, Jin H, Wang M, Hu Y, Chen S, He Q, Chang J, Hong C, Zhou Y, Wang D, Miao X, Li Y, Hu B. Neurologic Manifestations of Hospitalized Patients With Coronavirus Disease 2019 in Wuhan, China. JAMA Neurol. 2020 Jun 1;77(6):683-690. doi: 10.1001/jamaneurol.2020.1127. PMID 32275288
- [Background] Boldrini P, Bernetti A, Fiore P; SIMFER Executive Committee, SIMFER Committee for International Affairs. Impact of COVID-19 outbreak on rehabilitation services and Physical and Rehabilitation Medicine physicians' activities in Italy. An official document of the Italian PRM Society (SIMFER). Eur J Phys Rehabil Med. 2020 Jun;56(3):316-318. doi: 10.23736/S1973-9087.20.06256-5. Epub 2020 Mar 16. No abstract available. PMID 32175719
- [Background] Griffiths J, Hatch RA, Bishop J, Morgan K, Jenkinson C, Cuthbertson BH, Brett SJ. An exploration of social and economic outcome and associated health-related quality of life after critical illness in general intensive care unit survivors: a 12-month follow-up study. Crit Care. 2013 May 28;17(3):R100. doi: 10.1186/cc12745. PMID 23714692
- [Background] Torres J, Carvalho D, Molinos E, Vales C, Ferreira A, Dias CC, Araujo R, Gomes E. The impact of the patient post-intensive care syndrome components upon caregiver burden. Med Intensiva. 2017 Nov;41(8):454-460. doi: 10.1016/j.medin.2016.12.005. Epub 2017 Feb 8. English, Spanish. PMID 28188064
- [Background] Elliott D, Davidson JE, Harvey MA, Bemis-Dougherty A, Hopkins RO, Iwashyna TJ, Wagner J, Weinert C, Wunsch H, Bienvenu OJ, Black G, Brady S, Brodsky MB, Deutschman C, Doepp D, Flatley C, Fosnight S, Gittler M, Gomez BT, Hyzy R, Louis D, Mandel R, Maxwell C, Muldoon SR, Perme CS, Reilly C, Robinson MR, Rubin E, Schmidt DM, Schuller J, Scruth E, Siegal E, Spill GR, Sprenger S, Straumanis JP, Sutton P, Swoboda SM, Twaddle ML, Needham DM. Exploring the scope of post-intensive care syndrome therapy and care: engagement of non-critical care providers and survivors in a second stakeholders meeting. Crit Care Med. 2014 Dec;42(12):2518-26. doi: 10.1097/CCM.0000000000000525. PMID 25083984
- [Background] Hayhurst CJ, Jackson JC, Archer KR, Thompson JL, Chandrasekhar R, Hughes CG. Pain and Its Long-term Interference of Daily Life After Critical Illness. Anesth Analg. 2018 Sep;127(3):690-697. doi: 10.1213/ANE.0000000000003358. PMID 29649027
- [Background] Battle CE, Lovett S, Hutchings H. Chronic pain in survivors of critical illness: a retrospective analysis of incidence and risk factors. Crit Care. 2013 May 29;17(3):R101. doi: 10.1186/cc12746. PMID 23718685
- [Derived] Ojeda A, Cunat T, Comino-Trinidad O, Aliaga J, Arias M, Calvo A. New-onset chronic and neuropathic pain in survivors of severe COVID-19: A secondary analysis of the PAIN-COVID Trial. Rev Esp Anestesiol Reanim (Engl Ed). 2025 Dec;72(10):501915. doi: 10.1016/j.redare.2025.501915. Epub 2025 Sep 23. PMID 40998165
- [Derived] Ojeda A, Calvo A, Cunat T, Mellado-Artigas R, Costas-Carrera A, Sanchez-Rodriguez MM, Comino-Trinidad O, Aliaga J, Arias M, Martinez-Palli G, Dursteler C, Ferrando C. Effectiveness of a specific follow up program for the management of the mental components of post-intensive care syndrome and chronic pain after COVID-19: results from the PAIN-COVID randomized clinical trial. Rev Esp Anestesiol Reanim (Engl Ed). 2024 May;71(5):349-359. doi: 10.1016/j.redare.2023.12.009. Epub 2024 Jan 17. PMID 38242358
- [Derived] Ojeda A, Calvo A, Cunat T, Mellado-Artigas R, Comino-Trinidad O, Aliaga J, Arias M, Ferrando C, Martinez-Palli G, Dursteler C. Characteristics and influence on quality of life of new-onset pain in critical COVID-19 survivors. Eur J Pain. 2022 Mar;26(3):680-694. doi: 10.1002/ejp.1897. Epub 2021 Dec 15. PMID 34866276
- [Derived] Ojeda A, Calvo A, Cunat T, Artigas RM, Comino-Trinidad O, Aliaga J, Arias M, Ahuir M, Ferrando C, Dursteler C. Rationale and study design of an early care, therapeutic education, and psychological intervention program for the management of post-intensive care syndrome and chronic pain after COVID-19 infection (PAIN-COVID): study protocol for a randomized controlled trial. Trials. 2021 Jul 24;22(1):486. doi: 10.1186/s13063-021-05463-7. PMID 34303381